CLINICAL TRIAL: NCT03724435
Title: ARRAY: Focused Ultrasound for the Treatment of PAncReatic CanceR - an InternAtional RegistrY
Brief Title: Focused Ultrasound for the Treatment of Pancreatic Cancer - an International Registry
Acronym: ARRAY
Status: Terminated | Type: Observational
Why Stopped: Competing trial will publish similar results
Sponsor: Focused Ultrasound Foundation (Other)
Collaborators: Navitas Clinical Research, Inc (Unknown)
Responsible Party: Sponsor
Other Study IDs: FUSREG001
Record Dates: First submitted 2018-08-31; First posted 2018-10-30 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Pancreatic Cancer
Keywords: pancreatic cancer; focused ultrasound
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Pancreatic Cancer Participants: No intervention will be administered. Assessments are performed as standard of care.

SUMMARY:
This pancreatic cancer registry aims to collect information on people around the world who select focused ultrasound (FUS) as part of their treatment for pancreatic cancer to learn about the performance of the focused ultrasound technology and health outcomes; the impact of focused ultrasound on your overall health; and provide an understanding of the current care for pancreatic cancer.

DETAILED DESCRIPTION:
The purpose of the registry is to collect data on the performance of the focused ultrasound (FUS) technology and health outcomes. A wide variety of approaches exist for using FUS on pancreatic cancer patients, and the primary goal is to capture this broad spectrum of approaches and their impact on patients overall health. This information will help provide a better understanding of current care, and may possibly direct further, more specific investigations that will follow this registry. After obtaining informed consent a baseline history, physical examination, laboratory studies, and imaging studies needed per standard of care will be performed. Patients' treatment is determined by their caregivers only, and thus the registry will evaluate patient management in "real-world" conditions.

Enrollment Goal: 100

Primary Outcomes: Pain related to pancreatic cancer, Objective response, Progression-free and overall survival, Performance Status, Clinical Benefit Response (CBR), Health-related quality of life

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Stated willingness to comply with all registry procedures and availability for the duration of the registry
* Histology proven pancreatic carcinoma in any area of pancreas
* Pancreatic tumor that can be treated by FUS
* Willingness and ability to complete follow-up interviews

Exclusion Criteria:

* Any disease, condition or surgery which would result in a contraindication to undergoing FUS therapy.
* Clinical trials of pancreatic cancer not of focused ultrasound or related activities
* Other non-pancreatic cancer clinical trials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The registry population will be drawn from patients who have been diagnosed with pancreatic cancer and are eligible for FUS therapy. Participants are allowed to receive standard-of-care treatment, including chemotherapy, radiation therapy, and best supportive care. Participants being treated in another FUS clinical trial may be included in this registry.
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2019-12-06 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Survival | 1 year
  Time until the occurence of death

OTHER OUTCOMES:
Pain Related to Pancreatic Cancer | Day 7, Day 14, Day 30, Day 60, Day 90, Every 90 days thereafter through survival, up to 36 months
  The proportion achieving a 2 point reduction or greater will be assessed at each time point and across time using the Brief Pain Inventory (Short Form). Pain will be rated from 0 (no pain) to 10 (pain as a bad as can imagine) .
Performance Status | Baseline, Day 30, Day 60, Day 90, Every 90 days thereafter through survival, up to 36 months
  Improvement in performance status for a period of at least 4 consecutive weeks without showing any sustained worsening.
Clinical Benefit Response (CBR) | Day 7, Day 14, Day 30, Day 60, Day 90, Every 90 days thereafter through survival, up to 36 months
  The proportion of participants with a CBR will be measured at each follow-up time point.
Impact on Quality of Life and Cost | Baseline, Day 1, Day 7, Day 14, Day 30, Day 60, Day 90, Every 90 days thereafter through survival, up to 36 months
  Standardized instrument to measure of health-related quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Joo Ha Hwang, MD, PhD, Principal Investigator — Stanford University; Joan Vidal-Jove, MD, PhD, Principal Investigator — Hospital Universitario Mútua Terrassa; Tim Meakem, MD, Study Director — Focused Ultrasound Foundation
Locations (4):
- Medical University of Pleven, Pleven, Bulgaria
- Seoul National University, Seoul, South Korea
- National Taiwan University Hospital, Taipei, Taiwan
- Oxford University Hospital, Headington, Oxford, United Kingdom